CLINICAL TRIAL: NCT03330574
Title: A Prospective, Longitudinal Study to Evaluate the Function of the Retina and Visual Pathways in Glaucoma Patients Using PERG
Brief Title: To Study the Function of the Retina in Glaucoma Patients Using PERG
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Swiss Vision Network (Other)
Responsible Party: Principal Investigator, Dr. Kaweh Mansouri, Doctor, Swiss Vision Network
Other Study IDs: PERG-01
Record Dates: First submitted 2017-10-12; First posted 2017-11-06 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Variability of the device: We will study the repeatability and reliability of the Diopsys® ERG Vision Testing Systems in normal non-glaucomatous people and in those with suspicion of glaucoma or confirmed glaucoma.
- Diagnosis and progression of glaucoma: Patients who have a suspicion of glaucoma and patients with confirmed glaucoma will be included. PERG data obtained by the Diopsys® ERG Vision Testing Systems will be analyzed to study the PERG changes in different clinical situations, such as early glaucoma and progression of glaucoma.
- Effect of medical/surgical intervention: Patients will undergo standard treatment based on their medical history and we will observe the PERG changes induced by these treatments (eye drops, laser or surgery) with the Diopsys® ERG Vision Testing Systems.

SUMMARY:
The purpose of this trial is to evaluate the performance of a new diagnostic device in the diagnosis and management of glaucoma. We will use this new device (PERG) to evaluate the function of the retina in glaucoma patients. This device is safe for the patients.

DETAILED DESCRIPTION:
Glaucoma is one of the leading causes of blindness worldwide. It's an optic neuropathy characterized by the progressive death of retinal ganglion cells.

In laboratories, it's possible to measure the electrical activity of retinal ganglion cells (RGC). Some researchers found that RGC showed electrical anomalies before dying. This decrease of electrical activity can be measured by using pattern electroretinography (PERG). Unfortunately, these measures could not be obtained in clinics before this new device.

For this reason, Diopsys developed a new device that can measure PERG directly in clinics, allowing physicians to have these data earlier to help them diagnose pathologies such as glaucoma or other ganglion cells abnormalities.

Currently, it is known that glaucoma is difficult to diagnose in the early stages and it's challenging to decide when to start a treatment.

In this study, our purpose is to use this new device to evaluate its efficacy in the diagnosis and management of glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma (all types of glaucoma);
* Ocular hypertensive (Suspicion of glaucoma);
* Control Patients (without any suspicion/sign of glaucoma);
* Have given written informed consent, prior to any investigational procedures;
* Aged 18 years of either sex.

Exclusion Criteria:

* Patients not able to understand the character of the study
* Participation in other clinical research within the last 4 weeks
* Other diseases that may cause visual field loss or optic disc abnormalities
* Systemic diseases that may affect PERG amplitude such as diabetes, parkinsonism, multiple sclerosis
* Poor best corrected visual acuity outside the limits recommended for the test
* Patients with high myopia (>5D)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients will be enrolled from glaucoma clinics of the Montchoisi glaucoma center
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Magnitude, μV | 4 years
  Strength of the signal
Magnitude D, μV | 4 years
  Strength and phase
MagD/Mag Ratio (no units) | 4 years
  Ratio between MagD and Mag
SNR, dB | 4 years
  Signal to Noise Ratio

CONTACTS AND LOCATIONS:
Overall Officials: Kaweh Mansouri, MD, Principal Investigator — Glaucoma Center, Montchoisi Clinic
Locations (1):
- Montchoisi Clinic, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No